CLINICAL TRIAL: NCT00219674
Title: Home Automatic External Defibrillator Training for High-Risk Patients
Brief Title: At-Home Automated External Defibrillator (AED) Training Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health - Seattle and King County (Other Government)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Susan Damon, Program Manager, Public Health - Seattle and King County
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01HL074098-01A1 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Myocardial Infarction; Heart Arrest; Chest Pain; Congestive Heart Failure; Angina, Unstable
Keywords: education; training, defibrillators; home defibrillators; automated external defibrillators; psychological adjustment
MeSH Terms: conditions — Myocardial Infarction; Heart Arrest; Chest Pain; Heart Failure; Angina, Unstable | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2 (Active Comparator): Group II
  Interventions: Behavioral: Group II: Video training + enhanced self-efficacy (SE)
- 3 (Active Comparator)
  Interventions: Behavioral: Group III: In-person training + enhanced SE
- 4 (Active Comparator)
  Interventions: Behavioral: Group IV: In-person training + enhanced SE + support
- 1 (Active Comparator): Group I
  Interventions: Behavioral: Group I: Video training

INTERVENTIONS:
Behavioral: Group I: Video training — Participants will receive the AED with a video that provides "instructional" training.
  Arms: 1
Behavioral: Group II: Video training + enhanced self-efficacy (SE) — Partcipants will receive the AED with instructional video, a manikin, and additional training materials by mail.
  Arms: 2
Behavioral: Group III: In-person training + enhanced SE — Participants will receive a face-to-face training session in their home as well as the AED with instructional video, manikin and training materials.
  Arms: 3
Behavioral: Group IV: In-person training + enhanced SE + support — Participants will receive a face-to-face training session in their home as well as the AED, instructional video, manikin, and a resource manual with information to enhance the family member's confidence in their role as care provider.
  Arms: 4

SUMMARY:
The purpose of the research is to determine the best automated external defibrillator (AED) training approach for high-risk patients and their family members with regard to AED skills retention and psychological adjustment.

DETAILED DESCRIPTION:
In the past 3 decades, advances in the understanding of the resuscitation of cardiac arrest have provided opportunities to strengthen the links in the chain of survival. Despite the apparent progress, however, survival has remained poor. Cardiac arrest is a leading cause of mortality in the US, accounting for up to 450,000 deaths annually. Eighty percent of all cardiac arrest events are caused by the arrhythmia, ventricular fibrillation. Prompt electrical defibrillation is the only effective therapy. The time interval from collapse to attempted defibrillation is the most important determinant of outcome. The chance of survival decreases on average by approximately 10-15% for every minute that elapses prior to attempted defibrillation. Thus, methods to decrease the time interval between collapse and electrical defibrillation represent a true opportunity to improve survival from cardiac arrest.

Even in communities where emergency medical systems are best situated to treat cardiac arrest, response intervals are on average greater than 6 minutes. The development of the automated external defibrillator (AED) provides the possibility to decrease the interval from collapse to defibrillation by enabling persons outside the traditional emergency medical services response system who are typically not trained in rhythm recognition to deliver life-saving therapy. The AED is a device that can be applied in case of cardiac arrest and will assess the heart rhythm and instruct the bystander whether to provide a shock. In addition, approximately 75% of cardiac arrests occur in the home and are witnessed or found by a family member. Thus, a family responder AED program, where family members of persons at relatively high risk of cardiac arrest are equipped and trained with AEDs, may in part, decrease the interval from collapse to shock in cardiac arrest and improve outcome. Persons who have recently been hospitalized for an acute coronary syndrome are known to be at elevated risk for cardiac arrest. Indeed, the provision of an AED for home use is already in practice. However, it is not clear what method should be used to train family members in this potentially lifesaving set of skills. The purpose of the proposed study is to evaluate 4 different AED training methods to determine if the training approaches differentially affect AED skill retention or psychological status. Although the programs span the spectrum from streamlined to personalized and intensive, each approach constitutes a potential real-world, generalizable AED training method.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for acute myocardial infarction, unstable angina, cardiac chest pain, congestive heart failure with ejection fraction less than 40, a cardiac procedure with a documented history of coronary artery disease
* Resides in Pierce, King, or Snohomish Counties, Washington (WA)
* Lives with someone physically and mentally able to operate an AED
* Able to provide written informed consent
* Has a telephone

Exclusion Criteria:

* Lives in a nursing home
* Do not resuscitate (DNR) orders checked on chart
* Suffers from a severe co-morbidity that prevents them from participating in a long-term study
* Has an implantable cardioverter defibrillator
* Non-English speaking patient and/or family member/significant other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2004-07; Primary Completion 2009-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
AED skills retention when assessed at 9 months from enrollment date | 9 months

SECONDARY OUTCOMES:
Psychological adjustment measured by a series of validated questionnaires administered at time of enrollment, 3 months, and 9 months | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Rea, MD, MPH, Principal Investigator — Division of Emergency Medical Services, Public Health - Seattle and King County
Locations (1):
- Division of Emergency Medical Services, Public Health - Seattle and King County, Seattle, Washington, United States

REFERENCES:
- [Derived] Meischke H, Diehr P, Phelps R, Damon S, Rea T. Psychologic effects of automated external defibrillator training: a randomized trial. Heart Lung. 2011 Nov-Dec;40(6):502-10. doi: 10.1016/j.hrtlng.2010.12.009. Epub 2011 Mar 16. PMID 21411144